CLINICAL TRIAL: NCT05732610
Title: MGC Health COVID-19 & Flu A+B Home Multi Test Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Group Care, LLC (Industry)
Collaborators: CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MGC-1001
Record Dates: First submitted 2023-02-15; First posted 2023-02-17 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Influenza A; Influenza B
Keywords: COVID-19; Flu A; Flu B; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Intervention Model Description: This is an open label study to evaluate the usability of the MGC Health COVID-19 & Flu A+B Home Multi Test using information from the Quick Reference Instructions (QRI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Individuals - ages 14 and older (Experimental): This test is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older.
  Interventions: Diagnostic Test: MGC Health COVID-19 & Flu A+B Home Multi Test
- Individuals - ages 2 to 13 (Experimental): This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples.
  If the subject is under the age of 14, an adult lay-user will collect the sample.
  Interventions: Diagnostic Test: MGC Health COVID-19 & Flu A+B Home Multi Test (2 to 13 y/o)

INTERVENTIONS:
Diagnostic Test: MGC Health COVID-19 & Flu A+B Home Multi Test — self-collected direct anterior nares swab samples
  Arms: Individuals - ages 14 and older
Diagnostic Test: MGC Health COVID-19 & Flu A+B Home Multi Test (2 to 13 y/o) — adult lay user collected anterior nares swab sample
  Arms: Individuals - ages 2 to 13

SUMMARY:
The purpose of this study is to evaluate the usability of the MGC Health COVID-19 & Flu A+B Home Multi Test in home use.

DETAILED DESCRIPTION:
The MGC Health COVID-19 & Flu A+B Home Multi Test is a lateral flow immunochromatographic antibody assay intended for the simultaneous qualitative detection and differentiation of the nucleocapsid antigen from SARS-CoV-2, influenza A and/or influenza B directly from anterior nasal swab specimens obtained from individuals, who are suspected of respiratory viral infection within five (5) days of symptom onset. This test is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older or adult lay user collected anterior nares swab samples from individuals aged 2 to 13 years.

The objective of the study is to determine the usability of the MGC Health COVID-19 & Flu A+B Home Multi Test in a simulated home use environment.

This is an open label study to evaluate the usability of the MGC Health COVID-19 & Flu A+B Home Multi Test using information from the Quick Reference Instructions (QRI).

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) approved informed consent / assent, if applicable, is signed and dated prior to any study related activities.
* Male and female subjects 2 years of age and older.
* Subject is willing to provide a self-collected nasal swab sample. (If the subject is under the age of 14, an adult lay user will collect the sample.)
* Subject agrees to complete all aspects of the study.

Exclusion Criteria:

* Subject has a visual impairment that cannot be restored with glasses or contact lenses.
* Subject has prior medical or laboratory training.
* Subject uses home diagnostics, e.g., glucose meters, HIV tests.
* Subject has prior knowledge of their current COVID-19 or flu infection status.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Cattano, RN, MSN, Study Director — CSSi LifeSciences
Locations (1):
- L&A Morales Healthcare, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four (34) subjects were screened and enrolled into the study. There were no screen failures or early terminations.
Groups:
- Individuals - Ages 2 to 13: This kit is intended for non-prescription home use with self-collected direct anterior nares swab samples.
  If the subject is under the age of 14, an adult lay-user will collect the sample.
  MGC Health COVID-19 & Flu A+B Home Multi Test (2 to 13 y/o): adult lay user collected anterior nares swab sample
Period: Overall Study
Arm/Group | Individuals - Ages 14 and Older | Individuals - Ages 2 to 13
Started | 19 | 15
Completed | 19 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usability Data Set: A total of 34 subjects were enrolled in the study. There were 15 subjects ranging in age from 2 to 13. The collection and result interpretation for these subjects under 14 were done by an adult lay user.
Arm/Group | Usability Data Set
Number analyzed (Participants) | 34
Age, Customized [Count of Participants; unit: Participants]
  < 14 years | 15
  ≥ 14 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34
Education [Count of Participants; unit: Participants]
  Pre-high school | 20
  High school graduate | 6
  Some college | 5
  College graduate | 3

OUTCOME MEASURES:

1. Primary Outcome: Usability of Quick Reference Instructions (QRI) - Critical Steps
Description: Assess the usability of the Quick Reference Instructions (QRI) based upon observer evaluation. The observer completed an observation form for each subject assessing whether the subject or adult lay user completed each critical task, and whether the task was performed correctly.
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Usability Data Set
Number analyzed (Participants) | 34
participants
  Swab each nostril, rotating swab against nostril at least 5 times. | 34
  Rotate nasal swab in sample collection tube liquid at least 5 times. | 34
  Lift swab out of the liquid in collection tube and squeeze the tube against the swab tip 3 times. | 34
  Squeeze the sample collection tube while removing the nasal swab. | 34
  Press the nozzle lid firmly onto the sample collection tube. | 34
  Transfer 3 drops from the sample collection tube into the sample well of the test cartridge. | 34
  Do not move or lift the test cassette. | 34
  Read the results between 15 and 20 minutes. | 34

2. Primary Outcome: Usability of Test Kit
Description: Assess the usability of the kit for home use based upon subject evaluation. adult lay users filled out a questionnaire regarding the ease of understanding the instructions provided by the QRI for obtaining the sample, performing the test, and reading and interpreting the results, and the ease of completing each task.
  The subject or adult lay user used the following 5-digit score to answer the questions:
  1. Very easy to understand
  2. Fairly easy to understand
  3. Easy
  4. Fairly difficult to understand
  5. Very Difficult
Time Frame: one hour
Measure: Mean (Full Range); unit: Mean score on a scale
Arm/Group | Usability Data Set
Number analyzed (Participants) | 34
Mean score on a scale
  Overall, how easy or difficult was it to understand the instructions to conduct the test? | 1.50 [1 to 3]
  How easy or difficult was it to open the test cassette package? | 1.62 [1 to 3]
  How easy or difficult was it to remove the sealed film covering from the sample collection tube? | 1.62 [1 to 3]
  How easy was it to understand how to collect the sample from your nose or from another person? | 1.71 [1 to 3]
  How easy or difficult was it to understand the instructions to swirl the swab in the collection tube | 1.53 [1 to 3]
  How easy was it understand how to lift the swab out of the liquid and squeeze in the collection tube | 1.47 [1 to 3]
  How easy or difficult was it to insert the nozzle lid onto the sample collection tube? | 1.32 [1 to 3]
  How easy was it to understand to add the sample from the collection tube to the sample well | 1.24 [1 to 3]
  How easy or difficult was it to add the 3 drops into the test cassette? | 1.24 [1 to 3]
  How easy or difficult was it to read the test results? | 1.26 [1 to 3]
  How easy was it to understand the instructions on how to interpret the results of the test? | 1.24 [1 to 3]

3. Primary Outcome: Usability of Quick Reference Instructions (QRI) - Subject Test Result and Observer Confirmation
Description: Assess the usability of the QRI based upon observer evaluation.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Usability Data Set
Number analyzed (Participants) | 34
Participants
  Negative | 15
  Positive Flu A | 6
  Positive Flu B | 2
  Positive COVID-19 | 11

4. Primary Outcome: Usability of Quick Reference Instructions (QRI) - Interpretation of Example Test Results
Description: Assess the usability of the QRI. Subjects or adult lay users were presented with 10 sample images of test results: 1 negative test, 7 positive tests, and 2 invalid tests.
Time Frame: 1 hour
Measure: Number; unit: Participants with correct interpretation
Groups:
- Usability Data Set: A total of 34 subjects were enrolled in the study. The collection and result interpretation for these subjects under 14 were done by an adult lay user.
Arm/Group | Usability Data Set
Number analyzed (Participants) | 34
Participants with correct interpretation
  Image 1 - invalid test (no lines) | 34
  Image 2 - positive Flu A | 34
  Image 3 - positive COVID-19, Flu A, and Flu B | 34
  Image 4 - invalid test (Flu A line, no C line) | 34
  Image 5 - positive Flu B | 33
  Image 6 - positive Flu A, and Flu B | 32
  Image 7 - negative | 34
  Image 8 - positive COVID-19 and Flu A | 19
  Image 9 - positive COVID-19 and Flu B | 31
  Image 10 - positive COVID-19 | 34

ADVERSE EVENTS:
Time Frame: 24 hours
Description: This study was deemed to have a less than significant risk by IRB assessment, and no sites reported any adverse events during or after the study enrollment period.
Arm/Group | Usability Data Set
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05732610/Prot_SAP_000.pdf